CLINICAL TRIAL: NCT02306915
Title: A Randomized, Double-Blind Study to Assess the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Single Subcutaneous Administration of Lipegfilgrastim (Doses up to 100 μg/kg) in Healthy Japanese and Caucasian Subjects
Brief Title: PK, PD, Safety and Tolerability of Lipegfilgrastim in Healthy Japanese and Caucasian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merckle GmbH (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: XM22-PK-10036
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Pharmacokinetics; Pharmacodynamics
Keywords: Lipegfilgrastim, Lonquex, Japanese Bridging
MeSH Terms: interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- lipegfilgrastim 30 (Experimental)
  Interventions: Drug: lipegfilgrastim
- lipegfilgrastim 60 (Experimental)
  Interventions: Drug: lipegfilgrastim
- lipegfilgrastim 100 (Experimental)
  Interventions: Drug: lipegfilgrastim

INTERVENTIONS:
Drug: lipegfilgrastim — lipegfilgrastim 30 μg/kg, 60 μg/kg, 100 μg/kg

SUMMARY:
Cohorts of Japanese participants will be enrolled and treated prior to cohorts of Caucasian participants for the sake of matching. Every effort will be made to match Caucasian and Japanese participants on a cohort basis at enrollment. Reasonable effort will be made to maintain balance between male and female participants within the cohorts. There will be no replacement of participants following randomization.

DETAILED DESCRIPTION:
Eligible participants will be admitted to the investigational center and after confirming their eligibility will be randomized to receive a single dose of 30, 60, or 100 μg/kg lipegfilgrastim. There will be 11 visits to the investigational center during the study, including a screening visit, 1 inpatient period (through Day 4 post-dose) and 9 ambulatory visits.

Blood samples for PK, PD and immunogenicity analysis will be collected pre-dose and at specified time points post-dose. A mandatory blood sample for pharmacogenetics (PGx) will be collected from all participants. During the study the following safety assessments will be performed: vital signs measurements,physical examinations, record of adverse events, clinical laboratory tests, urinalysis, safety ECG recordings, local tolerability (injection site reactions), overall tolerability, pregnancy testing, spleen sonography, and concomitant medications

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18.0 and ≤25 kg/m2.
* Body weight must be ≥ 50 kg and ≤ 90 kg.
* Is in good general health as determined by medical history, physical examination, 12-lead electrocardiography (ECG), vital signs and clinical laboratory tests.
* Subjects are able to read, write and understand English or Japanese; they must be able to understand the requirements of the study and be willing to comply with all trial requirements.
* Female subjects of childbearing potential must have a negative serum β-human chorionic gonadotropin (β-hCG) test at screening and negative urine pregnancy test at check-in. All subjects must be either surgically sterile (for females that means documented complete hysterectomy, bilateral oophorectomyor bi-tubal ligations; partial hysterectomy is not sufficient), abstinent throughout the study or, if of reproductive capacity and not abstinent, exercising any 2 different forms of highly effective contraception methods with his/her partner during the entire study period.

  o Additional inclusion criteria for Japanese subjects:
* Subject must be a non-naturalized Japanese citizen and hold a Japanese passport.
* Subject must have/had 2 Japanese parents and 4 Japanese grandparents who are all non-naturalized Japanese citizens, as confirmed by interview.
* Subject has been living outside of Japan for 10 years or fewer as confirmed by interview.

  o Additional inclusion criterion for Caucasian subjects:
* The subject is Caucasian, and confirms by interview that his/her parents and grandparents are Caucasian and none are of Black/African descent, Middle-Eastern descent or Asian descent.
* -other criteria apply, please contact the investigator for more information

Exclusion Criteria:

* History of hypersensitivity to pegfilgrastim, filgrastim, lenograstim, Escherichia coli derived proteins, or to any excipients (glacial acetic acid, sodium hydroxide, sorbitol, polysorbate 20).
* Prior exposure to filgrastim, pegfilgrastim or lenograstim or other granulocyte colony stimulating factors (G-CSFs) in clinical development less than 6 months before randomization.
* Findings of splenomegaly on sonography, defined by splenic length in excess of 12.3 cm (Andrews, 2000; Benter et al, 2011) and clinical judgment.
* Existence or recent history of persistent pulmonary infiltrates or recent pneumonia, or current symptoms of upper respiratory infection. In the case of pneumonia, subject may be screened 12 weeks following cessation of antibiotic treatment.
* -other criteria apply, please contact the investigator for more information

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
PK: Area under the serum concentration-time curve (AUC), from time 0 to the last measurable concentration (AUC0-t) | Days 1-8, 10, 14, 17, 21
  2 hours for visits 3, 9; 1 day for visit 10
AUC from time 0 extrapolated to infinity (AUC0-∞) | Days 1-8, 10, 14, 17, 21
Maximum observed serum drug concentration (Cmax) | Days 1-8, 10, 14, 17, 21
Time to maximum observed serum drug concentration (tmax) | Days 1-8, 10, 14, 17, 21
The percentage of the extrapolated area to infinity in relation to the total area under the curve (%AUCext) | Visits 3, 9, 10
Apparent serum terminal elimination rate constant (λz) | Days 1-8, 10, 14, 17, 21
  2 hours for visits 3, 9; 1 day for visit 10
Associated elimination half-life (t½) | Days 1-8, 10, 14, 17, 21
Mean residence time (MRT) | Days 1-8, 10, 14, 17, 21
Apparent total body clearance (CL/F) | Days 1-8, 10, 14, 17, 21
Apparent volume of distribution during the terminal phase (Vz/F) | Days 1-8, 10, 14, 17, 21
PD: ANC area over baseline effect curve (ANC AOBEC) | Days 1-8, 10, 14, 17, 21
Maximum measured ANC value after dosing (ANC Cmax) | Days 1-8, 10, 14, 17, 21
Time point at which ANC Cmax is observed (ANC tmax) | Days 1-8, 10, 14, 17, 21
Time (days) until ANC returns to baseline value | Days 1-8, 10, 14, 17, 21
CD34+ area over the baseline effect curve (CD34+ AOBEC) | Days 1-8, 10, 14, 17, 21
Maximum measured CD34+ value after dosing (CD34+ Cmax) | Days 1-8, 10, 14, 17, 21
Time point at which CD34+ Cmax is observed (CD34+ tmax) | Days 1-8, 10, 14, 17, 21

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (1):
- Teva Investigational Site 34193, London, United Kingdom